CLINICAL TRIAL: NCT02689999
Title: The Effect of Dexrabeprazole on Intragastric and Intraesophageal Acidity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Neutec Ar-Ge San ve Tic A.Ş (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEU-01.15
Record Dates: First submitted 2016-02-10; First posted 2016-02-24 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: Gastroesophageal Reflux Disease (GERD), GERD, impedence
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dexrabeprazole 10 mg Enteric-Coated Tablets (Experimental): Dexrabeprazole 10 mg Enteric-Coated Tablets / once daily
  Interventions: Drug: Dexrabeprazole 10 mg Enteric-Coated Tablets

INTERVENTIONS:
Drug: Dexrabeprazole 10 mg Enteric-Coated Tablets

SUMMARY:
It is planned to investigate the effect of dexrabeprazole on gastric acid primarily, and then gastroesophageal reflux disease (GERD) symptoms, intraesophageal acidity (reflux) and impedance kinetics.

DETAILED DESCRIPTION:
The participants will be on one week medication after two-weeks observation period. Intragastric and intraesophageal multichannel intraluminal impedance-pH (pH-MII) monitoring will be performed before and after medication. The pre- and post-treatment data will be compared. The safety tests will be performed during study in terms of possible side effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of gastroesophageal reflux disease (GERD) in presence of pyrosis and/or regurgitation occurs once a week or more.
* Esophagitis stage A-B according to Los Angeles classification,
* Major symptom should be gastroesophageal reflux disease (GERD) in presence of overlapping symptoms,
* Age range should be 18-70 years,
* BMI should be 18-33 kg/m2,
* Presence of sufficient gastric acidity: Cases which intragastric ph > 4 value is under 25% according to dual multichannel intraluminal impedance-pH MII monitoring performed before study initiation,
* Pathologic intraesophageal acid exposure; DeMeester score > 14.75 and/or ph < 4 value > 4% (according to at 21 hour measurement at least),
* Helicobacter pylori should be negative according to biopsy in gastrointestinal system (GIS) endoscopy performed in last 12 months before study initiation; if biopsy not performed in endoscopy, stool antigen test or urease breath test should be performed and Helicobacter pylori should be negative.

Exclusion Criteria:

* Presence of food in stomach in gastrointestinal system (GIS) endoscopy performed in last 12 months before study initiation, all types of gastrointestinal system (GIS) pathology such as Barret stricture, stomach channel obstruction, malignity, gastrointestinal system (GIS) bleeding and cases with > 3 cm Hiatus hernia.
* Presence of severe chronic comorbid diseases; uncontrolled or insulin-dependent diabetes mellitus (IDDM), symptomatic gallbladder stone (cases who are asymptomatic and are not undergo cholecystitis and whose stone is 3 cm or polyp is smaller than 1 cm may be included), active or unhealed stomach or duodenum ulcer, Zollinger-Ellison syndrome, primary esophagus motility disorders, pancreatitis, inflammatory bowel disease, chronic liver disease, severe liver disease, uncontrolled renal impairment, presence of cancer except non-melanoma skin cancer, heart failure, cerebrovascular disease, epilepsy,
* Major psychiatric disease,
* Alcoholism or cases take narcotics,
* Pathologic laboratory test; hemogram, sedimentation, C-reactive protein (CRP), thyroid function tests, liver enzymes,
* Malabsorption that may affect drug absorption,
* Immunosuppressive and cortisone taking cases,
* Pregnancy or positive pregnancy test and lactating women,
* Cases taking all types of drugs which may affect gastrointestinal system motility or acid release,
* Cases undergo abdominal operation; hysterectomy, abdominal hernia operation, caesarean, appendectomies may be included but all types of cholecystectomy will be excluded.
* Cases taking a proton pomp inhibitor (PPI) and H2 blocker for last seven days and prokinetic drug for last three days,
* Condition that taking drugs need stomach acid for optimal absorption; such as ketoconazole, iron salts, digoxin, ampicillin esters, anticoagulants, antineoplastic agents.
* Cases who must take prostaglandin analogs,
* Cases who must take non-steroidal anti-inflammatory drug (NSAID) during study,
* Cases taking antidepressants,
* Cases who refuse to sign informed consent,
* Hypersensitivity to study drug.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-02; Primary Completion 2017-05 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
- The percent of pH < 4 duration of 24-hour intragastric acidity and intraesophageal acidity after seven-days treatment. | One week
  Multichannel intraluminal esophageal impedance pH-meter will be applied to cases in screening and second visit in order to evaluate the effect on 24-hour intragastric and intraesophageal acid values. 24-hour pH values of cases will be measured with pH-meter. Combined impedence pH catheter will be placed to 10 cm under and 5 cm upper of inferior esophageal sphincter of cases under local anesthesia. Cases will be informed about adherence to the diet list, not to take anti-acids and need to press symptom button on device when complaints occur during 24-hour measurements. After 24 hours, results will be recorded and reported by transferring to computer environment. These results will be compared with measurement obtained in screening visit and then efficacy assessment will be done.
- The area under curve (AUC) of pH < 4 duration of 24-hour intragastric acidity and intraesophageal acidity after seven-days treatment. | One week
  Multichannel intraluminal esophageal impedance pH-meter will be applied to cases in screening and second visit in order to evaluate the effect on 24-hour intragastric and intraesophageal acid values. 24-hour pH values of cases will be measured with pH-meter. Combined impedence pH catheter will be placed to 10 cm under and 5 cm upper of inferior esophageal sphincter of cases under local anesthesia. Cases will be informed about adherence to the diet list, not to take anti-acids and need to press symptom button on device when complaints occur during 24-hour measurements. After 24 hours, results will be recorded and reported by transferring to computer environment. These results will be compared with measurement obtained in screening visit and then efficacy assessment will be done.

CONTACTS AND LOCATIONS:
Locations (3):
- Turkey (Türkiye) (3):
  - Ege University Gastroenterology Department, Izmir, Bornova
  - Ankara University Gastroenterology Department, Ankara
  - On Dokuz Mayıs University Gastroenterology Department, Samsun

IPD SHARING:
Plan to Share IPD: Undecided